CLINICAL TRIAL: NCT00641992
Title: Prognosis Factors of the Response After Medical Treatment of Amebic Liver Abscess
Brief Title: Prognosis of Failure Treatment of Amebic Liver Abscess
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other); Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Dr. Martin Sanchez Aguilar, Epidemiologia Clinica, Universidad Autonoma de San Luis Potosí
Other Study IDs: PFP-ALA
Record Dates: First submitted 2008-03-12; First posted 2008-03-24 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Amebic Liver Abscess
Keywords: amebic liver abscess; failure; prognosis
MeSH Terms: conditions — Liver Abscess, Amebic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Response to medical treatment
- 2: Failure to medical treatment (surgery or percutaneous resolution)

SUMMARY:
Amebic liver abscess is the most frequent extra-intestinal form of the amoebiasis; actually the factors for predicting failure in the medical treatment are not clear. We conducted trial for determining the clinical value of paraclinical factor in this issue.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical, ultrasonographic and serologic diagnosis (ELISA) of amebic liver abscess.
2. Both genders
3. Older 15 years

Exclusion Criteria:

1. Clinically suspected piogenous liver abscess
2. Positive hemoculture
3. Negative ELISA for amoebic antigens
4. Immunosupresion (HIV)
5. Abdominal or biliary surgery antecedents
6. Abdominal neoplasia antecedents

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: sequential patients with clinical, ultrasonographic and serologic diagnosis (ELISA) of amebic liver abscess
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 1999-05; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Failure of medical treatment | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Martín Sánchez-Aguilar 1, MSc, Principal Investigator — 1. Department of Experimental Surgery, Faculty of Medicine, Universidad Autónoma de San Luis Potosí; Onofre Morán-Mendoza, PhD, Study Director — Department of Clinical Epidemiology, Faculty of Medicine, Universidad Autónoma de San Luis Potosí
Locations (2):
- Mexico (2):
  - Department of Surgery, Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán"., Mexico City, Mexico DF
  - Faculty of Medicine, Universidad Autónoma de San Luis Potosí, San Luis Potosí City, San Luis Potosí